CLINICAL TRIAL: NCT04388423
Title: Study on Application of Simulated Training in Ultrasound Guided Transversus Abdominis Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yi Liu, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PLAGHAOC202003
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Transversus Abdominis Plane Block; Simulation Training; Learning Curve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental)
  Interventions: Other: simulated puncture training
- Group C (Experimental)
  Interventions: Other: traditional bedside teaching

INTERVENTIONS:
Other: simulated puncture training — The residents are trained of simulated puncture : 1.the location puncture; 2. finding fixed-point needle on the model for 5 times, each time for 30 minutes.
  Arms: Group S
Other: traditional bedside teaching — The residents are trained by traditional bedside teaching
  Arms: Group C

SUMMARY:
With the development of society and the enhancement of people's awareness of law and self-protection, it is necessary to use simulation technology to create a simulated human and clinical environment to replace the traditional teaching of clinical operation on real patients. So simulation teaching is more and more important in medical education. However, simulation teaching is in the ascendant in China, especially in the ultrasound-guided nerve block, limited by the lack of full simulation of puncture model, the simulation training of ultrasound-guided nerve block is not carried out much. Therefore, this study uses simulation training to carry out ultrasound-guided horizontal abdominal muscle block teaching, in order to explore an effective way of ultrasound-guided nerve block teaching.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old; ASA 1 ~ 2; patients under non-transvaginal gynecologic surgery, rectal surgery or descending colon surgery

Exclusion Criteria:

* Patients with communication disorder Central or peripheral nervous system diseases. Liver and kidney functions seriously damaged Coagulation function abnormality and local anesthetic allergy history Patients with serious heart disease, hypertension and diabetes. Patients who have used analgesic drugs or drugs that may affect cardiovascular function within 24 hours before operation.

Patients with infection at the puncture site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
The time taken to complete the blocking operation | procedure/surgery
  After finishing the disinfection sheet, the operator began to perform unilateral transversal muscle planar ultrasound scanning, positioning and puncture until the end of injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Haidian, China